CLINICAL TRIAL: NCT00119119
Title: Efficacy and Safety of the Association With Pentoxyphilline and Tocopherol on the Fibrosis in Patients With Chronic Hepatitis C
Brief Title: Efficacy and Safety of Pentoxyphilline and Tocopherol on the Fibrosis in Patients With Chronic Hepatitis C
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: French National Agency for Research on AIDS and Viral Hepatitis (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ANRSHC10 PENTO
Record Dates: First submitted 2005-07-04; First posted 2005-07-13 (Estimated); Last update posted 2007-01-12 (Estimated); Status verified 2007-01

CONDITIONS: Hepatitis C, Chronic; Liver Fibrosis
Keywords: Hepatitis C; Liver Cirrhosis; Tocopherols
MeSH Terms: conditions — Hepatitis C, Chronic; Liver Cirrhosis; Hepatitis C | interventions — Tocopherols

INTERVENTIONS:
Drug: pentoxyphilline
Drug: tocopherol

SUMMARY:
The fibrosis of liver is a complication of chronic hepatitis C. There is actually no established treatment for fibrosis of the liver. Pentoxyphilline and tocopherol may have an activity on fibrosis. The aim of the study is to analyse the efficacy and the safety of the combination with pentoxyphilline and tocopherol (12 months) on liver fibrosis, in patients with chronic hepatitis C, who are non-long-term responders, or with intolerance or contra-indication to interferon-alfa and ribavirin.

DETAILED DESCRIPTION:
The aim of this study is to analyse the efficacy and the safety of the combination of pentoxyphilline (400 mg, twice a day) and tocopherol (500 mg, twice a day), given during 12 months on the fibrosis related to HCV chronic hepatitis in 100 patients who are non-long-term responders, or with contra-indication or intolerance to the current treatment of reference (combination with interferon-alfa and ribavirin). It is a therapeutic, national, multicentric, double-blind, placebo-controlled phase III trial. The patients included had histological liver injuries with a Metavir score of A 0 to 2, F 2 or 3 and no other etiology of liver disease. The primary objective is to analyse the variation of the liver fibrosis evaluated by morphometric analysis between the 2 liver biopsies performed at the end of the trial and within 3 years before the treatment. The secondary objectives are the variation of the Metavir fibrosis and activity scores, of serum markers of fibrosis (hyaluronate, PIIIP, TNF-alfa, fibrotest) and ALT between the end and the beginning of the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 75 years
* Chronic hepatitis C defined by positive HCV Ab and HCV RNA and histological proven injuries
* Liver biopsy with a size over or equal to 15mm, performed within 3 years of enrolment, with a Metavir score of activity from 0 to 2 and fibrosis score of 2 or 3.
* Non long term responders or patients with contra-indication or intolerance to interferon alfa or ribavirin
* No anti-viral treatment during the trial
* Signed written informed consent

Exclusion Criteria:

* Alcohol consumption over or equal to 40 g/d
* Allergy to tocopherol or pentoxyphilline
* Treatment with platelet anti-aggregates, anti-vitamin K, theophylline, armophylline
* Treatment with tocopherol or pentoxyphilline since the last liver biopsy
* Pregnancy, breast feeding, lack of contraception
* Decompensated cirrhosis, organ graft, chronic renal insufficiency
* BMI over 27
* Diabetes type I or II
* Other etiology of liver disease (HBV, HIV, hemochromatosis, alfa-1 antitrypsin deficiency, Wilson's disease, auto-immune hepatitis, drug-related hepatitis)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2002-02; Study Completion 2006-12

PRIMARY OUTCOMES:
Variation of the percentage of liver fibrosis evaluated with morphometric analysis between the liver biopsies performed at the end and before the trial (defined as significant if over 5 percent).

SECONDARY OUTCOMES:
Variation of fibrosis Metavir score between the two biopsies
Variation of activity Metavir score between the two biopsies
Variation of liver markers of fibrosis : hyaluronate, N-terminal peptide of procollagen III, TNF-alfa and fibrotest
Variation of ALT

CONTACTS AND LOCATIONS:
Overall Officials: Helene Fontaine, MD, Principal Investigator — Service d'hepatologie Hopital Necker Paris
Locations (1):
- Service d'hepatologie Hopital Necker, Paris, France